CLINICAL TRIAL: NCT06144294
Title: Whole-Body Hyperthermia for Mood and Anxiety Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-01025619
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Depression; Mood Disorders; Anxiety Disorders; Postpartum Anxiety
Keywords: postpartum depression; mood disorders; anxiety disorders; postpartum anxiety; whole-body hyperthermia; antidepressant therapy; anxiolytic therapy; postpartum feasibility and acceptability; psychoneuroimmunology; Broad-band neural suppression; EEG; Likert scale; inflammatory activity; pro-inflammatory cytokines; precision functional brain maps; fMRI
MeSH Terms: conditions — Depression, Postpartum; Mood Disorders; Anxiety Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group 2 - Cohort 2a (Experimental): Healthy women or transgender men 18-50 years of age, <6 months postpartum
  Interventions: Other: Whole-Body Hyperthermia
- Group 2 - Cohort 2b (Experimental): Women and transgender men 18-50 years of age, <6 months postpartum, meeting criteria for a major depressive episode in the postpartum period on the MINI
  Interventions: Other: Whole-Body Hyperthermia
- Group 2 - Cohort 2c (Experimental): Healthy adults of both sexes 18-50 years of age
  Interventions: Other: Whole-Body Hyperthermia
- Group 2 - Cohort 2d (Experimental): Adults of both sexes 18-50 years of age meeting criteria for an episode of major depression or generalized anxiety disorder on the MINI
  Interventions: Other: Whole-Body Hyperthermia
- Group 3 - Cohort 2a (Experimental): Healthy women or transgender men 18-50 years of age, <6 months postpartum
  Interventions: Other: Whole-Body Hyperthermia; Diagnostic Test: fMRI
- Group 3 - Cohort 2b (Experimental): Women and transgender men 18-50 years of age, <6 months postpartum, meeting criteria for a major depressive episode in the postpartum period on the MINI
  Interventions: Other: Whole-Body Hyperthermia; Diagnostic Test: fMRI
- Group 3 - Cohort 2c (Experimental): Healthy adults of both sexes 18-50 years of age
  Interventions: Other: Whole-Body Hyperthermia; Diagnostic Test: fMRI
- Group 3 - Cohort 2d (Experimental): Adults of both sexes 18-50 years of age meeting criteria for an episode of major depression or generalized anxiety disorder on the MINI
  Interventions: Other: Whole-Body Hyperthermia; Diagnostic Test: fMRI

INTERVENTIONS:
Other: Whole-Body Hyperthermia — The Clearlight dome sauna is portable infrared sauna consisting of two lightweight domes and an infrared heating pad. The sauna will be used to deliver the intervention to the participant and the sauna session will end as soon as (1) an internal body temperature of 38.5 C (101.3 F) is reached for two consecutive minutes or, (2) 140 minutes have passed.
  Other Names: Clearlight Portable Dome Sauna
Diagnostic Test: fMRI — A standard magnetic resonance imaging (fMRI) machine will be used to take images of the brain.
  Arms: Group 3 - Cohort 2a; Group 3 - Cohort 2b; Group 3 - Cohort 2c; Group 3 - Cohort 2d

SUMMARY:
This study aims to examine the scientific mechanisms of whole-body hyperthermia (WBH), a novel, rapidly acting, single session antidepressant and anxiolytic therapy. It also aims to determine its feasibility and acceptability in women with postpartum depression (PPD). The study will enroll four cohorts of participants: healthy postpartum controls; postpartum women with PPD; healthy adult controls; and adults with major depressive disorder or anxiety disorders in a longitudinal protocol.

DETAILED DESCRIPTION:
Whole-body hyperthermia has already been shown to be feasible, acceptable, and effective in major depressive disorder (MDD) populations, with an open-label study and a subsequent randomized, double-blind, sham-controlled study both demonstrating efficacy. Some evidence indicates that the antidepressant effect may be due to immune mechanisms, though it may also be mediated through direct neural effects of hyperthermia

This project aims to establish a protocol to deliver WBH therapy to patients with mood and anxiety disorders to collect information about scientific mechanisms. It also seeks to extend treatment to a specific population: a single session WBH treatment could be of tremendous interest to depressed postpartum women who wish to avoid medications and time away from their infants.

The mechanistic work will be completed with the four cohorts. By examining mechanisms in all four groups, investigators will be able to determine mechanisms unique to ill individuals as well as any mechanistic differences between MDD and PPD. In addition, the investigators aim to establish feasibility and acceptability of this protocol in postpartum women. Why? Over 80% of women deliver a child, and 15-20% of all women develop significant postpartum mental illness, usually depression and anxiety.

Participants will be divided into two groups: those undergoing a simplified protocol to test feasibility and acceptability in the postpartum (Study Group 1) and those undergoing a more time-intensive protocol to evaluate mechanisms (Study Group 2). In addition, participants in Study Group 2 will be eligible to enroll in a sub-study (Study Group 3) including up to 10 fMRI session.

ELIGIBILITY:
Inclusion Criteria

* Study Group 2

  * Arm 1: Healthy women or transgender men 18-50 years of age, ≤ 6 months postpartum
  * Arm 2: Women and transgender men 18-50 years of age, ≤ 6 months postpartum, meeting criteria for a major depressive episode in the postpartum period on the MINI.
  * Arm 3: Healthy adults of both sexes 18-50 years of age.
  * Arm 4: Adults of both sexes 18-50 years of age meeting criteria for an episode of major depression or generalized anxiety disorder on the Mini International Neuropsychiatric Interview (MINI)
* Study Group 3

  * Subjects enrolled in Study Group 2 are eligible for an optional additional sub-study (Study Group 3); inclusion criteria are the same as for Study Group 2.

Exclusion criteria for all:

* For logistics, we will exclude individuals with BMI >30 and waist size > 35, who may not fit comfortably in the sauna dome for all cohorts described above.
* For contraindications to hyperthermia, we will exclude from all cohorts listed above, individuals with severe cardiovascular disease, including congestive heart failure, coronary artery disease, uncontrolled hypertension, and hypotension; pregnancy; active substance use disorders; recent major injuries or surgeries (<1 week prior); impaired sweating (those with multiple sclerosis, diabetes mellitus with neuropathy, central nervous system disease, heat insensitivity); a history or family history of malignant hyperthermia, fever or active signs of infection; taking medications that may have interactions with hyperthermia (for example, barbiturates, diuretics, and beta blockers) and the use of an antipyretic or anihistamine medication in the 12 hours prior to the WBH intervention. Individuals with above mentioned conditions will be excluded since either WBH might deteriorate their conditions or it is unknown how their condition will be affected by WBH.
* For contraindications to immune analyses, we will exclude individuals with conditions that might affect immune analyses, including individuals with known active autoimmune or endocrine disease and individuals with active infection at baseline.

Additional exclusion criteria by cohort or applicable study group:

* Study Group 2

  * Arm 1: For psychiatric contraindications, we will exclude individuals with a history of psychiatric disorders as assessed by MINI since the cohort will consist of mentally healthy individuals as a control group.
  * Arm 2: For psychiatric contraindications, we will exclude individuals with bipolar disorder or other Axis I psychiatric disorders except depressive and anxiety disorders and individuals taking antidepressants who are unwilling to hold antidepressant dose steady from recruitment through study termination. In this cohort we exclude individuals with other psychiatric disorders except depressive and anxiety disorders to rule out the effect of other psychiatric diseases on the outcome.
  * Arm 3: For psychiatric contraindications, we will exclude individuals with a history of psychiatric disorders as assessed by MINI since the cohort will consist of mentally healthy individuals as a control group.
  * Arm 4: For psychiatric contraindications, we will exclude individuals with bipolar disorder or other Axis I psychiatric disorders except depressive and anxiety disorders and individuals taking antidepressants who are unwilling to hold antidepressant dose steady from recruitment through study termination. In this cohort we exclude individuals with other psychiatric disorders except depressive and anxiety disorders to rule out the effect of other psychiatric diseases on the outcome.
* Study Group 2 and Study Group 3 - All participants

  * For contraindications to use of the e-Celsius capsule that will be used to measure core temperature, we will exclude individuals with pacemakers or any other electric medical implant, individuals with a current intestinal disorder that could lead to obstruction of the digestive tract including gastroparesis, individuals with history of diverticula, individuals with history of past surgical procedures in the gastrointestinal tract, individuals with a swallowing disorder and individuals with Crohn's disease.
* Study Group 3 - All participants

  * For contraindications to MRI, individuals with metal in the body will be excluded from participating in the MRI portion of the research since magnetic fields in MRI scanners can cause dangerous interactions in patients with metallic foreign bodies: projectile effect, twisting, burning, artifacts, and device malfunction (interference with a pacemaker).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Percent change in EEG amplitude. | During the course of the intervention: when participant core temperature reaches 38.5 C for two consecutive minutes OR after 140 minutes have passed.
  Measure the extent of broad-band neural suppression in WBH.
Percent change in EEG frequency. | During the course of the intervention: when participant core temperature reaches 38.5 C for two consecutive minutes OR after 140 minutes have passed.
  Measure the extent of broad-band neural suppression in WBH,

SECONDARY OUTCOMES:
Mean change from baseline in inflammatory activity as measured by pro-inflammatory cytokines. | Two days prior to the intervention; immediately prior to intervention; immediately post-intervention; and at five days post-intervention.
  Determine whether peripheral immune activation predicts the effect of WBH on PPD or depressive and anxiety symptoms in non-postpartum adults.
Mean change in average 24-hour core temperature. | Two days prior to the intervention and five days post-intervention.
  Determine the average change in core temperature across the whole-body hyperthermia intervention.
Individualized precision functional brain maps. | Up to 3 fMRI scans in the 10 days before the intervention and up to 7 fMRI scans in the 6 weeks post-intervention.
  Determine longitudinal changes in neural circuit activity produced by whole-body hyperthermia.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Osborne, PhD, Principal Investigator — Weill Medical College of Cornell University; Jonathan Power, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabral R, Prior PF, Scott DF, Brierley JB. Reversible profound depression of cerebral electrical activity in hyperthermia. Electroencephalogr Clin Neurophysiol. 1977 May;42(5):697-701. doi: 10.1016/0013-4694(77)90286-3. PMID 67029
- [Background] de Labra C, Pardo-Vazquez JL, Cudeiro J, Rivadulla C. Hyperthermia-Induced Changes in EEG of Anesthetized Mice Subjected to Passive Heat Exposure. Front Syst Neurosci. 2021 Sep 9;15:709337. doi: 10.3389/fnsys.2021.709337. eCollection 2021. PMID 34566589
- [Background] Yamane T, Tateishi A, Cho S, Manabe S, Yamanashi M, Dezawa A, Yasukouchi H, Ishioka K. The effects of hyperthermia on the spinal cord. Spine (Phila Pa 1976). 1992 Nov;17(11):1386-91. doi: 10.1097/00007632-199211000-00020. PMID 1462216
- [Background] Haveman J, Geerdink AG, Rodermond HM. Cytokine production after whole body and localized hyperthermia. Int J Hyperthermia. 1996 Nov-Dec;12(6):791-800. doi: 10.3109/02656739609027685. PMID 8950159
- [Background] Landsberg L, Young JB, Leonard WR, Linsenmeier RA, Turek FW. Is obesity associated with lower body temperatures? Core temperature: a forgotten variable in energy balance. Metabolism. 2009 Jun;58(6):871-6. doi: 10.1016/j.metabol.2009.02.017. PMID 19375759
- [Background] Lynch CJ, Power JD, Scult MA, Dubin M, Gunning FM, Liston C. Rapid Precision Functional Mapping of Individuals Using Multi-Echo fMRI. Cell Rep. 2020 Dec 22;33(12):108540. doi: 10.1016/j.celrep.2020.108540. PMID 33357444
- [Background] Newbold DJ, Laumann TO, Hoyt CR, Hampton JM, Montez DF, Raut RV, Ortega M, Mitra A, Nielsen AN, Miller DB, Adeyemo B, Nguyen AL, Scheidter KM, Tanenbaum AB, Van AN, Marek S, Schlaggar BL, Carter AR, Greene DJ, Gordon EM, Raichle ME, Petersen SE, Snyder AZ, Dosenbach NUF. Plasticity and Spontaneous Activity Pulses in Disused Human Brain Circuits. Neuron. 2020 Aug 5;107(3):580-589.e6. doi: 10.1016/j.neuron.2020.05.007. Epub 2020 Jun 16. PMID 32778224
- [Background] Mason AE, Fisher SM, Chowdhary A, Guvva E, Veasna D, Floyd E, Fender SB, Raison C. Feasibility and acceptability of a Whole-Body hyperthermia (WBH) protocol. Int J Hyperthermia. 2021;38(1):1529-1535. doi: 10.1080/02656736.2021.1991010. PMID 34674592
- [Background] Lindahl V, Pearson JL, Colpe L. Prevalence of suicidality during pregnancy and the postpartum. Arch Womens Ment Health. 2005 Jun;8(2):77-87. doi: 10.1007/s00737-005-0080-1. Epub 2005 May 11. PMID 15883651
- [Background] Maternal depression and child development. Paediatr Child Health. 2004 Oct;9(8):575-598. doi: 10.1093/pch/9.8.575. No abstract available. PMID 19680490
- [Background] Feldman R, Granat A, Pariente C, Kanety H, Kuint J, Gilboa-Schechtman E. Maternal depression and anxiety across the postpartum year and infant social engagement, fear regulation, and stress reactivity. J Am Acad Child Adolesc Psychiatry. 2009 Sep;48(9):919-927. doi: 10.1097/CHI.0b013e3181b21651. PMID 19625979
- [Background] Halligan SL, Murray L, Martins C, Cooper PJ. Maternal depression and psychiatric outcomes in adolescent offspring: a 13-year longitudinal study. J Affect Disord. 2007 Jan;97(1-3):145-54. doi: 10.1016/j.jad.2006.06.010. Epub 2006 Jul 24. PMID 16863660
- [Background] Lyons-Ruth K, Zoll D, Connell D, Grunebaum HU. The depressed mother and her one-year-old infant: environment, interaction, attachment, and infant development. New Dir Child Dev. 1986 Winter;(34):61-82. doi: 10.1002/cd.23219863407. No abstract available. PMID 3822211
- [Background] Murray L. The impact of postnatal depression on infant development. J Child Psychol Psychiatry. 1992 Mar;33(3):543-61. doi: 10.1111/j.1469-7610.1992.tb00890.x. PMID 1577898
- [Background] Righetti-Veltema M, Conne-Perreard E, Bousquet A, Manzano J. Postpartum depression and mother-infant relationship at 3 months old. J Affect Disord. 2002 Aug;70(3):291-306. doi: 10.1016/s0165-0327(01)00367-6. PMID 12128241
- [Background] Righetti-Veltema M, Bousquet A, Manzano J. Impact of postpartum depressive symptoms on mother and her 18-month-old infant. Eur Child Adolesc Psychiatry. 2003 Apr;12(2):75-83. doi: 10.1007/s00787-003-0311-9. PMID 12664271
- [Background] Field T. Postpartum depression effects on early interactions, parenting, and safety practices: a review. Infant Behav Dev. 2010 Feb;33(1):1-6. doi: 10.1016/j.infbeh.2009.10.005. Epub 2009 Dec 3. PMID 19962196
- [Background] McEvoy K, Osborne LM, Nanavati J, Payne JL. Reproductive Affective Disorders: a Review of the Genetic Evidence for Premenstrual Dysphoric Disorder and Postpartum Depression. Curr Psychiatry Rep. 2017 Oct 30;19(12):94. doi: 10.1007/s11920-017-0852-0. PMID 29082433
- [Background] Weissman MM. Postpartum Depression and Its Long-term Impact on Children: Many New Questions. JAMA Psychiatry. 2018 Mar 1;75(3):227-228. doi: 10.1001/jamapsychiatry.2017.4265. No abstract available. PMID 29387871
- [Background] Societal Costs of Untreated Perinatal Mood and Anxiety Disorders in the United States. Mathematica. Accessed December 1, 2022. https://www.mathematica.org/publications/societal-costs-of-untreated-perinatal-moodand- anxiety-disorders-in-the-united-states
- [Background] Cox EQ, Sowa NA, Meltzer-Brody SE, Gaynes BN. The Perinatal Depression Treatment Cascade: Baby Steps Toward Improving Outcomes. J Clin Psychiatry. 2016 Sep;77(9):1189-1200. doi: 10.4088/JCP.15r10174. PMID 27780317
- [Background] Koltyn KF, Robins HI, Schmitt CL, Cohen JD, Morgan WP. Changes in mood state following whole-body hyperthermia. Int J Hyperthermia. 1992 May-Jun;8(3):305-7. doi: 10.3109/02656739209021785. PMID 1607735
- [Background] LEHMANN HE. Combined pharmaco-fever treatment with imipramine (tofranil) and typhoid vaccine in the management of depressive conditions. Am J Psychiatry. 1960 Oct;117:356-8. doi: 10.1176/ajp.117.4.356. No abstract available. PMID 13760463
- [Background] Zschaeck S, Weingartner J, Ghadjar P, Wust P, Mehrhof F, Kalinauskaite G, Ehrhardt VH, Hartmann V, Tinhofer I, Heiland M, Coordes A, Kofla G, Budach V, Stromberger C, Beck M. Fever range whole body hyperthermia for re-irradiation of head and neck squamous cell carcinomas: Final results of a prospective study. Oral Oncol. 2021 May;116:105240. doi: 10.1016/j.oraloncology.2021.105240. Epub 2021 Feb 21. PMID 33626457
- [Background] Hanusch KU, Janssen CH, Billheimer D, Jenkins I, Spurgeon E, Lowry CA, Raison CL. Whole-body hyperthermia for the treatment of major depression: associations with thermoregulatory cooling. Am J Psychiatry. 2013 Jul;170(7):802-4. doi: 10.1176/appi.ajp.2013.12111395. No abstract available. PMID 23820835
- [Background] Janssen CW, Lowry CA, Mehl MR, Allen JJ, Kelly KL, Gartner DE, Medrano A, Begay TK, Rentscher K, White JJ, Fridman A, Roberts LJ, Robbins ML, Hanusch KU, Cole SP, Raison CL. Whole-Body Hyperthermia for the Treatment of Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Aug 1;73(8):789-95. doi: 10.1001/jamapsychiatry.2016.1031. PMID 27172277
- See also: Clearlight Sauna Dome — http://infraredsauna.com/curve-sauna-dome/